CLINICAL TRIAL: NCT00687492
Title: Centralized Pan-Asian Survey on the Under Treatment of Hypercholesterolemia
Acronym: CEPHEUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Joher Raniwalla, AstraZeneca
Other Study IDs: NIS-CAP-DUM-2008/1
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; NCEP ATP III guidelines; survey
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The survey will try to establish the proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the third NCEP ATP guidelines, overall and by country.

ELIGIBILITY:
Inclusion Criteria:

* 2 or more risk factors (according to NCEP ATP III guideline)
* Receiving lipid-lowering drug treatment for at least 3 months without dosage change for a minimum of 6 weeks.

Exclusion Criteria:

* Involvement in the planning and conduct of the study (applies to both AstraZeneca staff or staff at the study site).
* Previous enrolment or randomisation of treatment in the present study.
* Participation in a clinical study during the last 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had to be on a lipid-lowering drug treatment for at least 3 months, with no dose change for a minimum of 6 weeks.
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The number and percentage of subjects achieving the LDL-C goals according to updated 2004 NCEP ATP Ⅲ guidelines(overall and by country) | After collecting all Patient Record Form.

SECONDARY OUTCOMES:
The number and percentage of subjects achieving the LDL-C goals according to the updated 2004 NCEP ATP Ⅲ guidelines for several subject subsets. | After collecting all Patient Record Form.
The association between achievement of LDL-C goals,according to the updated 2004 NCEP ATPⅢ guidelines and patient and physician variables. | After collecting all Patient Record Form.
The physician characteristics associated with the allocation of hypercholesterolemia treatment regime. | After collecting all Patient Record Form.

CONTACTS AND LOCATIONS:
Overall Officials: Park Jeong Euy, Principal Investigator — Sungkyunkwan University
Locations (59):
- Research Site, Hong Kong, Hong Kong, China
- Indonesia (6):
  - Research Site, Semarang, Central Java
  - Research Site, Jakarta, DKI Jakarta
  - Research Site, Sidoarjo, East Java
  - Research Site, Surabaya, East Java
  - Research Site, Medan, North Sumatra
  - Research Site, Bandung, West Java
- Malaysia (19):
  - Research Site, Bangsar, Kuala Lumpur
  - Research Site, Kepong, Kuala Lumpur
  - Research Site, Kuala Lumpur, Kuala Lumpur
  - Research Site, Puchong, Kuala Lumpur
  - Research Site, Setapak, Kuala Lumpur
  - Research Site, Ampang, Selangor
  - Research Site, Batu Caves, Selangor
  - Research Site, Hulu Selangor, Selangor
  - Research Site, Kampung Baru Subang, Selangor
  - Research Site, Klang, Selangor
  - Research Site, Kuala Selangor, Selangor
  - Research Site, Petaling Jaya, Selangor
  - Research Site, Port Klang, Selangor
  - Research Site, Sekinchan, Selangor
  - Research Site, Seri Kembangan, Selangor
  - Research Site, Shah Alam, Selangor
  - Research Site, Subang Jaya, Selangor
  - Research Site, Sungai Buloh, Selangor
  - Research Site, Sunway City, Selangor
- Philippines (5):
  - Research Site, Lipa, Batangas
  - Research Site, Baguio City, Benguet
  - Research Site, Davao City, Davao Region
  - Research Site, Iloilo City, Iloilo
  - Research Site, Manila, Manila
- South Korea (15):
  - Research Site, Cheonan, Chung-Cheong-nam-do
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Bundang, Gyeonggi-do
  - Research Site, Guri-si, Gyeonggi-do
  - Research Site, Il-san, Gyeonggi-do
  - Research Site, Suwon, Gyeonggi-do
  - Research Site, Masan, Gyung-sang-nam-do
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Jeju City
  - Research Site, Seoul
  - Research Site, Ulsan
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (6):
  - Research Site, Bangkoknoi, Bangkok
  - Research Site, Dusit, Bangkok
  - Research Site, Pathumwan, Bangkok
  - Research Site, Ratchathewi, Bangkok
  - Research Site, Klongluang, Changwat Pathum Thani
  - Research Site, Muang, ChiangMai
- Vietnam (2):
  - Research Site, Hanoi, Hanoi
  - Research Site, Ho Chi Minh City, Hcmc